CLINICAL TRIAL: NCT05332002
Title: A Phase II Study of sFOLFOXIRI in Advanced Gastroesophageal Cancer (SAGE)
Brief Title: sFOLFOXIRI in Advanced Gastroesophageal Cancer, (SAGE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Patrick M Boland, MD, Assistant Professor, Rutgers Cancer Institute of New Jersey, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072204; Pro2022000268 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2022-03-29; First posted 2022-04-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Gastro-Intestinal Cancer
Keywords: Gastric and esophageal cancers (GEC)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4week alternating FOLFOX and a combination chemotherapy regime FOLFIRI (sFOLFOXIRI), (Other): A cycle will constitute 28 days of treatment, which will consist of one chemotherapy combination, either FOLFOX or FOLFIRI as below:
  1. Odd Cycles (e.g. 1, 3, 5, etc…) - mFOLFOX6 initiated on days 1 & 15: (Oxaliplatin 85 mg/m2 IV, leucovorin 400 mg/m2, 5FU 400 mg/m2 bolus, then 5FU 2400 mg/m2 over 46 hours)
  2. Even Cycles (e.g. 2,4,6, etc…) - FOLFIRI initiated on days 1 & 15: (Irinotecan 180 mg/m2 IV, leucovorin 400 mg/m2, 5FU 400 mg/m2 bolus, then 5FU 2400 mg/m2 over 46 hours)
  3. Nivolumab (optional, in-line with labelled approval) - 240 mg every 2 weeks
  Interventions: Drug: Four week alternating FOLFOX and FOLFIRI (sFOLFOXIRI)

INTERVENTIONS:
Drug: Four week alternating FOLFOX and FOLFIRI (sFOLFOXIRI) — This is a Single Arm Phase II trial of q4week alternating FOLFOX and FOLFIRI (sFOLFOXIRI), with or without nivolumab, in advanced human epidermal growth factor receptor 2 (HER2) negative gastric and esophageal cancers (GEC).
  The study treatment is a chemotherapy combination of either FOLFOX or FOLFIRI as below:
  1. mFOLFOX6: (Oxaliplatin 85 mg/m2 IV, leucovorin 400 mg/m2, 5-FU 400 mg/m2 bolus, then 5-FU 2400 mg/m2:
  2. FOLFIRI: (Irinotecan 180 mg/m2 IV, leucovorin 400 mg/m2, 5-FU 400 mg/m2 bolus, then 5-FU 2400 mg/m2
  3. Nivolumab(Optional) The chemotherapy combination of FOLFOX and FOLFIRI is a FDA approved treatment for advanced bowel and gastric

SUMMARY:
The primary objective is to determine the clinical efficacy of treatment regimen in terms of objective response rate (ORR). The secondary objectives is to determine the clinical efficacy of the study treatment in terms of progression free survival (PFS) and overall survival (OS). Additionally, to characterize the safety and toxicity profile of the study treatment as measured by the adverse event rates.

DETAILED DESCRIPTION:
The overall purpose of this protocol is to serve as a Single Arm Phase II trial of a four week alternating FOLFOX and FOLFIRI (sFOLFOXIRI), with or without nivolumab, in advanced human epidermal growth factor receptor two (HER2) negative gastric and esophageal cancers (GEC). This study evaluates the hypothesis that the use of sFOLFOXIRI in gastroesophageal cancer (GEC) will increase response rates beyond that expected with FOLFOX, while maintaining acceptable tolerability. The primary endpoint of this study is the objective response rate (ORR) while the key secondary endpoints include the progression free survival (PFS), overall survival (OS), and adverse event (AE) rates. The goal of this study is to establish the activity level of sFOLFOXIRI, with the thought that this could be further developed in the metastatic and/or peri-operative space if a sufficiently interesting degree of efficacy is observed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed metastatic or unresectable adenocarcinoma of esophageal, gastroesophageal junction or gastric origin
* Tumor is HER2 negative by standard local testing methodology
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 - 2
* Measurable disease by response evaluation criteria in solid tumors (RECIST) v1.1
* No prior systemic therapy for the present cancer given in the metastatic setting and > 6 months from administration of peri-operative chemotherapy, if applicable

  o Note: up to two prior cycles of mFOLFOX6 for the present illness is permitted if patients otherwise qualify for the study with adequate baseline imaging
* At least 18 years of age
* Adequate bone marrow and organ functions as defined by:
* Absolute neutrophil count ≥ 1500 cells/ μL
* Hemoglobin ≥ 8 g/ dL
* Platelets > 100,000 / μL
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance ≥ 30 mL/min by Cockroft-Gault
* Total bilirubin ≤ ULN
* Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) < 2.5 x ULN, unless with liver metastases and then must be <5 x ULN of normal
* Women and men of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect pregnancy on study, she must notify her treating physician immediately.
* Ability to understand the nature of this study protocol and give written informed consent.
* Willingness and ability to comply with scheduled visits, treatment plans laboratory tests and other study procedures.

Exclusion Criteria:

* Receipt of any investigational agents at the time of registration
* Known, untreated brain metastases
* Grade two or greater peripheral neuropathy
* Presence of any additional active malignancy within the past three years where the malignancy is at least reasonably likely to later the course of therapy, require systemic therapy or interfere with imaging assessments
* For those patients who are going to receive nivolumab
* No active use of systemic corticosteroids at the time of enrollment, at a dose equivalent of 10 mg/day or prednisone
* Clinically significant autoimmune disease which is active or has required systemic immunosuppression within the last two years
* Prior organ transplant or bone marrow transplant
* History of interstitial lung disease or pneumonitis
* Uncontrolled intercurrent illness, including significant active infection, symptomatic congestive heart failure, unstable angina or active arrhythmia
* Major surgery within the four weeks prior to initiation of study treatment
* A history of allergy or hypersensitivity to any of the study drugs
* Any additional significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from fully participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors ( RECIST) criteria version 1.1 | Three Years
  To determine the clinical efficacy of treatment regimen in terms of objective response rate.
Progression Free Survival (PFS) | Three Years
  To determine the clinical efficacy of the study treatment in terms of progressive free survival.
Overall Survival (OS) | Three Years
  To determine the clinical efficacy of the study treatment in terms of overall survival.
Adverse Event Rates | Three Years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boland, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Brunswick, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No